CLINICAL TRIAL: NCT06557746
Title: Coca-Cola Versus Supplemental Oxygen on Fatigue Management in Tibet Surgeons
Brief Title: Coca-Cola vs. Oxygen for Fatigue Management in Tibet Surgeons
Acronym: COMETS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Tibet Autonomous Region People's Hospital (Other)
Responsible Party: Principal Investigator, DONG WU, Professor of Gastroenterology, Tibet Autonomous Region People's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ME-TBHP-24-019
Record Dates: First submitted 2024-08-03; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Fatigue
Keywords: Surgeon Fatigue; Supplemental oxygen; Coca-Cola
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized controlled trial
Masking Description: Due to the nature of the intervention and the outcome measurement methods, it is difficult to blind both the participants and outcome assessors in this study. The investigators estimate that the impact of knowing the intervention group should be minimal, because the measurement of the outcomes in this study is relatively objective.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cola group (Experimental): 100 ml cola every 30 minutes during the operation
  Interventions: Other: Coca-Cola
- Oxygen group (Experimental): Continuous supply of oxygen (2 L/min) during the operation
  Interventions: Other: Supplemental oxygen

INTERVENTIONS:
Other: Coca-Cola — 100 ml Coca-Cola every 30 minutes during the operation
  Arms: Cola group
Other: Supplemental oxygen — Continuous supply of oxygen (2 L/min) during the operation
  Arms: Oxygen group

SUMMARY:
The study will be conducted among surgeons in Tibet, comparing the effects of Coca-Cola and supplemental oxygen on fatigue alleviation. Additionally, pre-planned subgroup analyses will examine the potential differences in effectiveness between Tibetan surgeons who have long lived in high-altitude areas and Han surgeons who work in these areas for shorter periods. The investigators hypothesize that for Tibetan surgeons, Coca-Cola will be more effective in alleviating fatigue, while for Han Chinese surgeons, supplemental oxygen will be more effective.

DETAILED DESCRIPTION:
Fatigue in surgeons can result in reduced concentration and muscle strength, compromising the safety of surgical procedures, particularly in high-altitude areas. In Tibet, surgeons often drink cola or inhale oxygen during operations, as these are believed to help alleviate fatigue. This study aims to evaluate the effects of Coca-Cola and supplemental oxygen in relieving fatigue among surgeons in Tibet and to investigate whether these effects vary based on the ethnicity of the doctors.

This study employs a stepped-wedge cluster randomized controlled trial design, recruiting 22 surgeons (k=22). Each doctor is scheduled to perform 24 surgeries and evaluated. At the beginning of the trial, all surgeons will drink cola. The supplemental oxygen will be administered in a random sequence to all participants until each has received the intervention. The primary outcome measure is the change in concentration performance scores before and after surgery (ΔCP). The secondary outcome measure is the change in maximum voluntary hand grip strength before and after surgery (ΔMVC). The study follows the intention-to-treat principle, including all subjects who have entered the randomization sequence in the analysis of the primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Surgeons employed at the People's Hospital of the Tibet Autonomous Region, including both Tibetan doctors with long-term experience in high-altitude areas and Han doctors working in high-altitude areas temporarily;
* Capable of serving as the lead surgeon in operations lasting at least 2 hours;
* Having lived and worked continuously in Lhasa for a minimum of 3 months, without traveling to low-altitude areas during this period;
* Fully understanding of this research and willing to sign a written informed consent form.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Attention decrease | 30 minutes before the surgery; end of the surgery; (the duration depends on the surgery complexity, at least 2 hours)
  Attention decrease is measured in terms of the difference in the concentration performance score (CP). The participants will take the d2 Test of Attention before and after every scheduled operation and get two CP scores (preoperative and postoperative). The higher the score, the better the attention. Therefore, a smaller difference (ΔCP) between preoperative and postoperative scores indicates a better effect in relieving fatigue.

SECONDARY OUTCOMES:
Maximal voluntary contraction force decrease | 30 minutes before the surgery; end of the surgery; (the duration depends on the surgery complexity, at least 2 hours)
  Maximal voluntary contraction force (MVC) is measured by hand dynamometer. The participants will be tested before and after every scheduled operation and get two MVC (preoperative and postoperative). The greater the strength, the less fatigued the hand muscles are. Therefore, a smaller difference (ΔMVC) between preoperative and postoperative scores indicates a better effect in relieving fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wu, M.D., Study Chair — Tibet Autonomous Region People's Hospital; Haifeng Xu, M.D., Study Chair — Tibet Autonomous Region People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dorion D, Darveau S. Do micropauses prevent surgeon's fatigue and loss of accuracy associated with prolonged surgery? An experimental prospective study. Ann Surg. 2013 Feb;257(2):256-9. doi: 10.1097/SLA.0b013e31825efe87. PMID 22824853